CLINICAL TRIAL: NCT01755832
Title: Better Everyday-life With Heated Pool Exercise Groups for Patients With Inflammatory Rheumatic Diseases
Brief Title: Heated Pool Exercise Groups for Patients With Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: National Resource Center for Rehabilitation in Rheumatology (Other)
Responsible Party: Principal Investigator, Anne Christie, Senior researcher, National Resource Center for Rehabilitation in Rheumatology
Other Study IDs: 2011/1654; NRF2012 (Other Grant/Funding Number: The Norwegian Rheumatism Association's Research Fund); OSL2012 (Other Grant/Funding Number: Oslo Sanitetsforenings Legater)
Record Dates: First submitted 2012-12-15; First posted 2012-12-24 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatic Disease
Keywords: inflammatory rheumatic joint disease; text message; > 18 years; Norwegian speaking
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pool exercise group: Patients with inflammatory rheumatic disease
  Interventions: Procedure: Pool exercise

INTERVENTIONS:
Procedure: Pool exercise — Group exercise in heated pool one hour per week for 12 weeks.

SUMMARY:
The purpose of this study is to investigate the effects of heated pool group exercises for patients with inflammatory rheumatic diseases with regard to symptoms (pain, fatigue, stiffness and ability to carry out daily activities).

DETAILED DESCRIPTION:
The patients receive text messages on mobile phones twice a week for circa 40 weeks. The text messages ask for pain, fatigue, stiffness and ability to carry out everyday activities. The patients should respond with a number from 0 to 10, where 0 is no symptoms/no hindering of activity and 10 is worst symptoms/worst hindering of activity.

ELIGIBILITY:
Inclusion Criteria:

* Referral from a medical doctor to group exercises in heated pool
* Inflammatory rheumatic joint disease
* > 18 years
* Stable disease
* Mobile phone owner
* Understand and use text messages on mobile phones

Exclusion Criteria:

* Independent living
* Joint surgery previous to the study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory rheumatic joint diseases with a medical referral to group exercises in heated pool.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Activity | 40 weeks
  How much do your health problems affect your ability to conduct daily activities? The outcome is assessed on a ten-point rating scale ranging from zero to ten with "0" representing "no affect" and "10" representing "extreme affect".
Pain | 40 weeks
  How much pain do you have at present? The outcome is measured on a ten-point numeric rating scale (NRS) ranging from zero to ten with "0" representing "no pain" and "10" representing "extreme pain".
Fatigue | 40 weeks
  How much fatigue do you have at present? The outcome is assesses on a ten-point rating scale ranging from zero to ten with "0" representing "no fatigue" and "10" representing "extreme fatigue"
Stiffness | 40 weeks
  How much stiffness do you have at present? The outcome is assessed on a ten-point numeric rating scale with "0" representing "no stiffness" and "10" representing "extreme stiffness".

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christie, Ph.D., Principal Investigator — National resource centre for rehabilitation in rheumatology
Locations (1):
- National resource center for rehabilitation in rheumatology, Oslo, Norway

REFERENCES:
- See also: Full text article — http://www.ncbi.nlm.nih.gov/pubmed/25490962